CLINICAL TRIAL: NCT06053073
Title: Induction to Labour With Double Cervical Ballon at Home Versus at Hospital to Improve the Vaginal Delivery Rate, Maternal Satisfaction and Reduce Costs: Multicentric Randomized Clinical Trial
Brief Title: Induction to Labour With Double Cervical Ballon at Home Versus at Hospital
Acronym: INDOBAMHOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-DBC-2021-35
Record Dates: First submitted 2023-09-06; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Induced; Birth; Cervical Dilatation; Live Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- At home patients group (Experimental): After insertion of the Cervical Rippening Balloon and checking fetal and maternal well-being, the patient will go home between 6 and 8 hours to complete the cervical rippening process. The patient will remove autonomously the balloon and will go to the hospital one hour later, where the induction will continue.
  Interventions: Device: Cervical rippening at home
- Hospitalized patients group (Active Comparator): After the insertion of the Cervical Rippening Balloon and verifications of the fetal and materna well-being, the patient will undergo the cervical rippening process for between 6 and 8 hours in the hospital and will remain hospitalized until the time of the delivery.
  Interventions: Device: Cervical rippening in the hospital

INTERVENTIONS:
Device: Cervical rippening at home — The experimental arm of the study will undergo cervical rippening at home between 6 and 8 hours and then will come back to the hospital to continue with the labor induction
  Arms: At home patients group
Device: Cervical rippening in the hospital — The active comparator arm of the study will undergo cervical rippening in the hospital between 6 and 8 hours and then will remain there to continue with the labor induction
  Arms: Hospitalized patients group

SUMMARY:
The goal of this clinical trial] is to compare the outcomes between induction to labour at home versus hospitalized. The main questions it aims to answer are:

* Can the induction to labour at home with cervical rippening ballon increase the vaginal delivery rate?
* Will the induction to labour at home increase maternal satisfaction
* Will the induction to labour at home improve medical circuits and coulb it be cost effective? Participants who meet inclusion criteria will undergo randomization so as to be asignated an induction to labour at home or in the hospital.

Researchers will compare both labour induction groups to see if the induction to labour at home has better outcomes as described previously.

DETAILED DESCRIPTION:
INDOBAMHOS is a multicentric randomized clinical trial which is based in the principle that cervical rippening with intracervical probes with ballons is as safe as pharmacological induction with PGE2 and it seems to be a suitable option to develop the cervical rippening process of the induction at home rather than in the hospital.

The purpouse of the study is to demonstrate that the comfort of performing the cervical rippenning at home will benefit patients with an increase of the vaginal delivery rate and increases maternal satisfaction. And also will improve medical circuits and could be cost-effective when compared to hospitalized labour induction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with ages >18 y.o
* Being able to read and understand the informed consent
* Accept to join the study when signing the informed consent
* Singleton
* Cephalic presentation
* Weeks of gestation between equal or more than 37 and less than 42
* Low risk indication of labor induction: Cronologically prolonged gestation
* Intermediate risk indication of labor induction: Macrosoma, Elevated maternal age, Intrahepatic Gestacional Colestasis, Gestational Diabetes Mellitus treated with diet, Gestational Diabetes Mellitus with insulin therapy and correct metabollic controls, Small for gestacional age fetus, Stable chronic hypertension, anterior caesarean section

Exclusion Criteria:

* Premature rupture of membranes (PROM)
* Breech presentation
* Unstable presentation
* Polihydramnios
* Severe congenital fetal afection
* Fetal growth restriction
* Suspected fetal well-being loss on CTG
* Bishop score equal or higher than seven before insertion of the CRB
* High cephalic presentation
* Home further than 30min from Hospital
* Preeclampsia
* Diabetes Mellitus type 1
* Maternal Hypertension
* Other maternal pathology with severe compromise
* Vaginal delivery Exclusion:
* Oclusive and non-occlusive placenta previa (marginal or low insertion)
* Vasa previa
* Transverse / Oblique situation
* Cord prolapse
* History of previous caesarean section with uterine incission in inverted T
* History of uterine rupture
* Two or more previous Caesarean section
* Active genital herpetical infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 834 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Type of delivery | End of the delivery
  Vaginal birth, Cesarean section

SECONDARY OUTCOMES:
Parity | At time of recruitment and end of delivery, about 1 or 2 days
  Number of pregnancies and deliveries of each patient
Indication of induction | 1 day
  Cathegorical variable, it will be studied the different reason that motivated the induction to delivery for each patient
Weeks of gestation | Only at time of recruitment, 1 day
  Measured in number of weeks and days
Bishop score | Before inserting the rippening balloon and after removing it, about 6 hours
  Score obtained when evaluating the different features of the uterine cervix by touch
Time of dilatation | During labour and until delivery, between 1 and 3 days
  Hours
Time of cervical rippening balloon | At the insertion of the rippening balloon and after removing it, about 6 hours
  Hours
Partian emptying of the balloon due to pain | During cervical rippening, about 6 hours
  Milliliters
Pharmacological analgesia during the cervical rippening | During cervical rippening, about 6 hours
  Number of drugs administered
Adverse outcomes | During cervical rippening and labor, between 6 hours and 3 days
  Number of adverse outcomes
Artificial Amniorrhexis | During cervical rippening and labor, between 6 hours and 3 days
  Presence or absence
Oxytocin infusion | During cervical rippening and labor, between 6 hours and 3 days
  Presence or absence
Subsequent PGE2 use | During cervical rippening and labor, between 6 hours and 3 days
  Presence or absence
Hyperstimulation | During cervical rippening and labor, between 6 hours and 3 days
  Presence or absence
Type of delivery | At the moment of the delivery, between 1 day and 3
  Cathegorical variable, it will be studied the different type of delivery for each patient
Time to delivery | At the moment of the delivery, between 1 day and 3
  Hours
Reason for instrumentation | At the moment of the delivery, between 1 day and 3
  Cathegorical variable, it will be studied the different reason of instrumentation
Reason for Cesarean section | At the moment of the delivery, between 1 day and 3
  Cathegorical variable, it will be studied the different reason of cesarean section
Epidural anesthesia | During cervical rippening and labor, between 6 hours and 3 days
  Presence of absence
Days of postpartum hospitalization | From the delivery to discharge from hospital, between 1 and 7 days
  Days
Fever during childbirth | At the moment of the delivery, between 1 day and 3
  Presence of absence
Perineal injuries | At the moment of the delivery, between 1 day and 3
  Presence of absence
Postpartum haemorrage | At the moment of the delivery, between 1 day and 3
  Presence of absence
Anemia | At the moment of the delivery, between 1 day and 3
  Presence of absence
Uterine rupture | At the moment of the delivery, between 1 day and 3
  Presence of absence
Maternal ICU admission | At the moment of the delivery, between 1 day and 3
  Presence of absence
Sepsis | At the moment of the delivery, between 1 day and 3
  Presence of absence
Meconial amniotic fluid | During cervical rippening and labor, between 6 hours and 3 days
  Presence of absence
Arterial pH | At the moment of the delivery, between 1 day and 3
  pH value of neonatal umbilical artery
Venous pH | At the moment of the delivery, between 1 day and 3
  pH value of neonatal umbilical vein
APGAR score | At the moment of the delivery, between 1 day and 3
  Score obtained when evaluating neonatal apearance, heart rate, muscular tone, activity, breath, gestures
Neonatal Intensive Care Unit (NICU) admission | From the delivery to discharge from hospital, between 1 and 7 days
  Days
Neonatal antibiotic administracion | From the delivery to discharge from hospital, between 1 and 7 days
  Presence of absence
Neonatal death | From the delivery to discharge from hospital, between 1 and 7 days
  Presence of absence
Hypoxic-ischemic encephalopathy | From the delivery to discharge from hospital, between 1 and 7 days
  Presence of absence
Neonatal seizures | From the delivery to discharge from hospital, between 1 and 7 days
  Presence of absence
Neonatal intubation or chest compressions | From the delivery to discharge from hospital, between 1 and 7 days
  Presence of absence
Persistent pulmonary hypertension of the newborn | From the delivery to discharge from hospital, between 1 and 7 days
  Presence of absence
Pain/Discomfort | During insertion of the cervical balloon, between 1 and 3 minutes
  Measure with analogue scale from 1 to 10
Pain/Discomfort | During cervical rippening, about 6 hours
  Measure with analogue scale from 1 to 10
Labor Agentry Scale | Up to two months
  Score obtained adding different items on the Scale
Edinburg questionnaire for postpartum depression | Up to two months
  Score obtained adding different items on the Scale
Impact of Event Scale-Revised | Up to two months
  Score obtained adding different items on the Scale
Breastfeeding | Up to two months
  Presence of abscence
SF-12 questionnaire | Up to two months
  Score obtained adding different items on the Scale
Diagnosis of depression | Up to two months
  Presence or Absence
Medical costs | One year
  Measured in euros

OTHER OUTCOMES:
Maternal age | At time of recruitment and end of delivery, about 1 or 2 days
  Years
Ethnicity | At time of recruitment and end of delivery, about 1 or 2 days
  Cathegorical variable, it will be studied the different ethnicities of the patients
Language spoken at home | At time of recruitment and end of delivery, about 1 or 2 days
  Cathegorical variable, it will be studied the different ethnicities of the patients
Socioeconomic data | At time of recruitment and end of delivery, about 1 or 2 days
  Number of people in the home, type of dwelling, socio-professional category, level of education
Height and weight | At time of recruitment and end of delivery, about 1 or 2 days
  Measured in centimeters and kilograms, combined in Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Llurba Olivé, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Maria del Carmen Medina Mallén, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Anna Mundó Fornell, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Ignacio Montoro Pacha, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Bruna Miarons Ferré, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Mitsury Flores, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rath W, Kehl S. The Renaissance of Transcervical Balloon Catheters for Cervical Ripening and Labour Induction. Geburtshilfe Frauenheilkd. 2015 Nov;75(11):1130-1139. doi: 10.1055/s-0035-1558094. PMID 26719596